CLINICAL TRIAL: NCT03058991
Title: Rescuing Cognitive and Emotional Regulatory Processes to Aid Smoking Prevention
Brief Title: Cognitive and Emotional Skills to Aid Smoking Prevention
Acronym: DOAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Claremont McKenna College (Other); Virginia Polytechnic Institute and State University (Other); Southern Methodist University (Other); University of Houston (Other)
Responsible Party: Principal Investigator, Michael Otto, Professor of Psychology, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21DA041531-01 (NIH); R21DA041531 (NIH)
Record Dates: First submitted 2016-10-07; First posted 2017-02-23 (Actual); Results first posted 2020-02-17 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Distress Tolerance Intervention (Experimental): For the Distress Tolerance Intervention, the investigators will use a Mindfulness Based Stress Reduction (MBSR) program that has been adapted for use with adolescents. This version of MBSR follows closely the original conceptualization developed by Kabat-Zinn. The focus is on formal and informal mindfulness practices, which encourage participants to foster intention, attention and attitude. The investigators will make slight modifications to the delivery of the MBSR intervention to take into account the developmental period of their participants (e.g., attention span) to encourage retention and increase relevancy. These changes will also allow the investigators to match the duration with their Working Memory Intervention.
  Interventions: Behavioral: Distress Tolerance Intervention
- Working Memory Intervention (Experimental): For the working memory training, the investigators will use the Cogmed RM program. Participants will be asked to use the program, while supervised twice a week, each time for an hour, for 8 weeks. Participants will also be asked to use the program on the other days for 25-35 minutes. The program resembles a video game, and comprises several different "games" that require visuo-spatial working memory (remembering the position of objects) and a combination of verbal and visual working memory (remembering phonemes, letters, and digits). The program adapts to the user's performance, such that trainees are able to perform at the limit of their ability, stimulating WM capacity adaptation.
  Interventions: Behavioral: Working Memory Intervention
- Control Informational Intervention (Active Comparator): This Control Informational Intervention has been used in the investigators' and other's previous studies. In the current application, it will match the session time of the Distress Tolerance and Working Memory interventions and will omit a focus on smoking (which is specific to the SPII intervention provided across all interventions), and will consist of discussions of a variety of healthy lifestyle topics, such as healthy eating, stress/time management, and recommended health screenings.
  Interventions: Behavioral: Control Informational Intervention

INTERVENTIONS:
Behavioral: Distress Tolerance Intervention — See arm/group description.
  Arms: Distress Tolerance Intervention
Behavioral: Working Memory Intervention — See arm/group description.
  Arms: Working Memory Intervention
Behavioral: Control Informational Intervention — See arm/group description.
  Arms: Control Informational Intervention

SUMMARY:
The purpose of the current proposal is to investigate the extent to which interventions designed to improve cognitive (working memory) and emotional (distress tolerance) regulatory processes enhance the effectiveness of standard no-smoking informational interventions. Emotional and cognitive dysregulation increases the likelihood of smoking and makes it particularly challenging to benefit from standard interventions. Working memory and associated deficits make it more difficult for individuals to utilize information from interventions, make judicious decisions regarding the cost and benefits of smoking, and to resist targeted advertising. In addition, disruptions in emotion regulatory capacities increase the probability of using cigarettes as a coping mechanism to self-regulate negative affect and stress. Individuals with affective disturbances smoke at higher rates and have more difficulties quitting, and are more likely to smoke as a way to reduce negative affect. The goal of the current project is to generate new insights and new approaches to smoking prevention among low-SES youth by investigating (1) the influence of known SES-related deficits in working memory and affect regulation on proximal measures of smoking risk, and (2) the potential for targeted interventions to reverse these risks. Specifically, the investigators examine the influence of working memory training and distress tolerance (mindfulness) interventions on cognitive/affective targets placing individuals at risk for smoking initiation and maintenance.

The specific aims of this study are therefore to investigate:

1. The feasibility and acceptability of school- and community-based brief interventions targeting working memory and distress tolerance in a diverse sample of low SES adolescents.
2. The effects of working memory and distress tolerance interventions, relative to a standard informational intervention alone, on specific cognitive-affective targets-delay discounting and distress tolerance--relevant to cigarette smoking initiation and maintenance.
3. The impact of cognitive /affective target activation on proximal measures of smoking risk/behavior and related health outcomes following intervention.

DETAILED DESCRIPTION:
Overview. The investigators are targeting a high-risk (low SES adolescents) population at a highly relevant period (high school) for smoking onset. The study design calls for block randomization of 150 non-smoking adolescents to one of three intervention conditions: (1) a control condition offering health education combined with a smoking prevention informational intervention (C+SPII), (2) a Working Memory intervention delivered prior to a smoking prevention informational intervention (WM+SPII), (3) a Distress Tolerance Intervention delivered prior to a smoking prevention informational intervention (DT+SPII). Smoking risk proximal outcomes are assessed by smoking propensity self-report, delay discounting, and implicit associations to smoking; smoking behavior is assessed at one-month follow-up.

Research material will consist of participant self-report of smoking, peer smoking, and parental smoking as well as self-report of personality characteristics (e.g. sensation seeking) that are associated with risk behaviors. Biological data (from exhalations) is also sampled for analysis of CO, to confirm non-smoking status.

Location of Interventions:

At this writing, the investigators are awaiting funding confirmation to decide among three options for how we will provide the interventions at the high school. The investigators have thought through and planned for the following three possibilities: (1) a school-time intervention in selected classroom space specific to the randomized intervention, (2) an afterschool intervention in open classroom space, and (3) an afterschool intervention in a community center. The investigators prefer these options in descending order (1 to 3), but final negotiation of space is pending their ability to confirm with the sites that the investigators will indeed do the project (have obtained funding). For example, as noted in the application, "the headmaster of Fenway High School, Peggy Kemp, is extremely supportive of our work, and plans to provide both institutional and social support in our endeavor." In the investigators' meetings with her, she suggested that the investigators try to provide the intervention during the school week; noting that these interventions fit the instructional demands for either the home room or PE time. Use of these in-school instructional slots would require approval of the school superintendent, but the process of obtaining such approval necessarily awaits confirmation of funding. The letters of support the investigators have obtained documents that if they are unable to realize option #1 or option #2, they can still realize this project demands by utilizing option #3.

Interventions: Participants will be randomized (using a random number table utilizing variable block sizes) to 1 of 3 study conditions according to two block randomization factors: sex and parental smoking status. Each intervention is to be delivered over eight consecutive weeks. Interventions are to be led by the Project Director, Dr. Eugenia Gorlin, with ongoing supervision from Drs. Otto and Doan. All interventions will be delivered in groups. Each of the study interventions is to be delivered twice a week over eight consecutive weeks. The school year for the targeted high school students lends itself to 8 waves of intervention. With 30 individuals per wave (randomized to 10 in each intervention for any given wave), the investigators anticipate achieving our full subject pool in 5 waves. Group nesting will be accounted for in the analytic plan.

The Smoking Prevention Informational Intervention (SPII) will be common to all randomized conditions in the study. The investigators selected the intervention from brief primary-care based interventions which followed the National Institutes of Health U.S. Public Health Service Tobacco Use and Dependence Clinical Practice Guideline. Youth will be provided with age-appropriate education on the norms and health consequences of smoking, affirmation of their non-smoking status, and help in developing a personalized strategy to maintain abstinence. Additionally, the investigators will incorporate a motivational interviewing component. Many of these elements are consistent with elements used in the youth MI program for adolescent smokers by Colby et al. (2005). The investigators will further incorporate into the SPII intervention Colby and associates' guided imagery about future smoking/non-smoking life status, and the initiation of our group sessions with open-ended exploration of the perceived likes and dislikes about smoking, and, during 4 sessions, provision of videotaped vignettes developed by the Massachusetts Department of Public Health to stimulate discussion on four content areas: health effects, social consequences, addiction, and financial cost. The SPII will be delivered following each of the 3 specific intervention conditions described in the "Study Arms" section.

All of the groups will have 8 weeks of training sessions, with sessions scheduled twice per week and each lasting up to 1 hour. Snacks will be served at these training sessions. In addition, participants will be asked to practice class skills (e.g., 20 min of practice 3 times a week) outside of these sessions for approximately 1 hour per week (for the memory program, this includes scheduling time in the computer room provided for this study).

Data Analysis Overview:

The following data analytic procedures are planned as of the current writing, but may be modified to incorporate new, more rigorous statistical modeling approaches as they become available.

1. The feasibility/ acceptability of school- and community-based brief interventions will be assessed by recruitment and attendance rates across the study period; acceptability (attendance of 80% of interventions by 70% of the randomized sample) will be assessed across the 3 conditions.
2. The investigators hypothesize that the WM+SPII and DT+SPII interventions, relative to C+SPII, will lead to higher WM and higher DT, respectively. Further, the investigators expect that WM will be higher in WM+SPII than in DT+SPII, and that DT will be higher in DT+SPII than in WM+SPII. The latter contrast will indicate if the two active treatments differ from each other on WM and/or DT; to perform these latter analyses, the investigators will replace the dummy variable contrasting WM+SPII and C+SPII, with a dummy variable comparing WM+SPII to DT+SPII.
3. To evaluate the impact of cognitive/affective target activation on proximal smoking risk/behavior following intervention, WM and DT will both be added (simultaneously) as time-varying predictors of outcome in MLM models for each of the 3 measures of smoking risk (susceptibility to smoking, implicit attitudes toward smoking, and delay discounting) and for actual smoking behavior (smoking behavior is dichotomous, so it will be analyzed using a GLMM with a logistic linking function). The regression coefficients for WM and DT predicting outcome in these models will indicate the degree to which each is related to smoking risk over and above the other, and controlling for the parallel change over time between these variables and the outcomes. This approach calculates the relation between both WN and DT with proximal measures of smoking risk within subjects over time. The Benjamini-Hochberg method will be used to correct for multiple statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (ages 12 years or older) enrolled in high school as a freshman or sophomore.
* Reflecting the demographics of the community in which we are recruiting, we expect approximately 70% of the sample to be at or below the poverty level, balanced between males and females, with the majority from an ethnic minority background.

Exclusion Criteria:

* Non-English speaking (operationalized as the inability to read and understand the consent form and converse in spoken English)

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Otto, Ph.D., Principal Investigator — Boston University; Stacey Doan, Ph.D., Principal Investigator — Claremont McKenna College
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Otto MW, Gorlin EI, Rosenfield D, Patten EA, Bickel WK, Zvolensky MJ, Doan SN. Rescuing cognitive and emotional regulatory skills to aid smoking prevention in at-risk youth: A randomized trial. Contemp Clin Trials. 2018 Jul;70:1-7. doi: 10.1016/j.cct.2018.04.005. Epub 2018 Apr 12. PMID 29655859
- [Background] Otto MW, Rosenfield D, Gorlin EI, Hoyt DL, Patten EA, Bickel WK, Zvolensky MJ, Doan SN. Targeting cognitive and emotional regulatory skills for smoking prevention in low-SES youth: A randomized trial of mindfulness and working memory interventions. Addict Behav. 2020 May;104:106262. doi: 10.1016/j.addbeh.2019.106262. Epub 2019 Dec 24. PMID 31918169

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 124 consented individuals, 108 were randomized and attended at least 1 session.
Groups:
- Working Memory Intervention: Participants were asked to use the CogMed RM program, while supervised twice a week, each time for an hour, for 8 weeks. Participants were also asked to use the program on the other days for 25-35 minutes. The program resembles a video game, and comprises several different "games" that require visuo-spatial working memory (remembering the position of objects) and a combination of verbal and visual working memory (remembering phonemes, letters, and digits). The program adapts to the user's performance, such that trainees are able to perform at the limit of their ability, stimulating WM capacity adaptation.
- Control Informational Intervention: This Control Informational Intervention has been used in the investigators' and other's previous studies. In this application, it matched the session time of the Distress Tolerance and Working Memory interventions and omitted a focus on smoking (which is specific to the SPII intervention provided across all interventions), and will consist of discussions of a variety of healthy lifestyle topics, such as healthy eating, stress/time management, and recommended health screenings.
- Distress Tolerance Intervention: For the Distress Tolerance Intervention, the investigators used a Mindfulness Based Stress Reduction (MBSR) program that has been adapted for use with adolescents. This version of MBSR follows closely the original conceptualization developed by Kabat-Zinn. The focus is on formal and informal mindfulness practices, which encourage participants to foster intention, attention and attitude. The investigators made slight modifications to the delivery of the MBSR intervention to take into account the developmental period of their participants (e.g., attention span) to encourage retention and increase relevancy. These changes allow the investigators to match the duration with their Working Memory Intervention.
Period: Overall Study
Arm/Group | Working Memory Intervention | Control Informational Intervention | Distress Tolerance Intervention
Started | 39 | 32 | 37
1-Week Follow Up | 23 | 27 | 28
Completed | 21 | 20 | 25
Not Completed | 18 | 12 | 12
Not completed — Lost to Follow-up | 17 | 12 | 12
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Working Memory Intervention | Control Informational Intervention | Distress Tolerance Intervention | Total
Number analyzed (Participants) | 39 | 32 | 37 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 32 | 37 | 108
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (1.3) | 14.2 (1.3) | 14.1 (1.2) | 14 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 20 | 59
  Male | 20 | 12 | 17 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 18 | 17 | 54
  Not Hispanic or Latino | 19 | 14 | 19 | 52
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 13 | 12 | 14 | 39
  Alaska Native or American Indian | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  White | 1 | 2 | 0 | 3
  Other | 21 | 16 | 18 | 55
  Decline to State | 0 | 1 | 2 | 3
  Multiracial | 0 | 0 | 0 | 0
  Unknown or Unreported | 2 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 39 | 32 | 37 | 108
Distress Tolerance [Mean (Standard Deviation); unit: z-score] — Distress Tolerance (DT) assessment includes the Distress Intolerance Index (DII) and the computerized Mirror-Tracing Persistence Task (MTPT-C) which are z-scored and aggregated to form a single DT index.The Distress Tolerance Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched children). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population and with higher scores reflecting worse tolerance. Population: Statistics are based on all cases with valid data for all variables in the model.
  z-score
    number analyzed (Participants) | 38 | 32 | 37 | 107
    (all) | .01 (.60) | -.01 (.76) | -.25 (.78) | -.09 (.72)
Smoking Susceptibility Assessment (SSA) [Mean (Standard Deviation); unit: Natural Log of Scores on a Scale] — Assessed with a 5-item scale asking about attitudes and likelihood of smoking with total scores ranging from 0 (no susceptibility) to 11 (highest susceptibility). The natural log of these scores are reported, with higher scores indicating higher susceptibility.
  Natural Log of Scores on a Scale | .23 (.51) | .29 (.49) | .43 (.57) | .31 (.53)
Smoking Brief Implicit Association Test (B-IAT) [Mean (Standard Deviation); unit: Standardized Difference Scores] — Participants sorted stimuli into "positive" or "negative" categories in 4 blocks--2 of which included "Smoking" and "I feel positive," the other 2 including "Smoking" and "I feel negative." Shorter response times when sorting "Smoking--Positive" versus "Smoking--Negative" blocks indicate implicit tendency to associate "smoking" with "positive." Standardized difference scores (d-scores) were computed using the improved scoring algorithm recommended by prior research (Greenwald, Banaji, & Nosek, 2003). Higher d-scores indicate less positive implicit attitudes towards smoking. Population: Statistics are based on all cases with valid data for all variables in the model.
  Standardized Difference Scores
    number analyzed (Participants) | 37 | 27 | 35 | 99
    (all) | .48 (.63) | .64 (.44) | .64 (.51) | .58 (.54)
Delay Discounting task [Mean (Standard Deviation); unit: Natural log of k-value] — Assessment includes a series of computerized decisions in which participants select a money award immediately or a larger award in 7, 14, or 30 days time. Participants were notified that they would be paid the amount selected on one randomly selected trial. K-values were submitted for analyses with higher scores representing great discounting of delayed rewards, meaning that higher scores reflect greater tendency to select the immediate award. Natural logs of K-values were used if K-values showed a large amount of skew. Population: Statistics are based on all cases with valid data for all variables in the model.
  Natural log of k-value
    number analyzed (Participants) | 38 | 32 | 37 | 107
    (all) | -2.9 (2.6) | -3.1 (1.9) | -2.7 (2.3) | -2.9 (2.3)
Work Memory Capacity [Mean (Standard Deviation); unit: z-score] — Assessment includes three computer-administered WM performance measures (N-back, Auditory Digit Span, and Corsi Block Tapping task) which are z-scored and aggregated to create a single WM index.The Working Memory Capacity Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched children). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population and higher scores reflecting greater capacity.
  z-score | -.16 (.62) | -.17 (.68) | .08 (.70) | -.08 (.67)
Actual Smoking Status [Mean (Standard Deviation); unit: Proportions of Smokers] — The piCO Smokerlyzer is a tool used to assess amount of carbon monoxide exhaled by a participant, with scores ranging from 0 to 150 parts per million (PPM), with scores under 3 indicating non-smoking and scores over 36 indicating very heavy addiction. The Timeline Follow Back is a self-report measure in which participants report the amount of cigarettes smoked each day for the last month. Mean proportions of smokers are reported (0=no smoking, 1=smoking) with smoking behaviors assessed via the piCO Smokerlyzer and the Timeline Follow Back. Population: Statistics are based on all cases with valid data for all variables in the model.
  Proportions of Smokers
    number analyzed (Participants) | 38 | 32 | 36 | 106
    (all) | .11 (.31) | .16 (.37) | .11 (.32) | .12 (.33)

OUTCOME MEASURES:

1. Primary Outcome: Specific Aim 1: Percentage of Participants Who Attended 13 or More Interventions
Description: Feasibility/acceptability of each intervention (indexed by attendance of at least 80% of interventions by 70% of the randomized sample) will be assessed.
Time Frame: Intervention (week 1 to week 8)
Population: Percentage of individuals who attended at least 80% of interventions reported.
Measure: Number; unit: percentage of participants
Arm/Group | Working Memory Intervention | Control Informational Intervention | Distress Tolerance Intervention
Number analyzed (Participants) | 39 | 32 | 37
percentage of participants | 41.0 | 50 | 40.5

2. Primary Outcome: Specific Aim 2: Working Memory Capacity
Description: Assessment includes three computer-administered WM performance measures (N-back, Auditory Digit Span, and Corsi Block Tapping task) which are z-scored and aggregated to create a single WM index.The Working Memory Capacity Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched children). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population and higher scores reflecting greater capacity.
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Working Memory Intervention | Control Informational Intervention | Distress Tolerance Intervention
Number analyzed (Participants) | 23 | 27 | 28
z-score | .06 (.86) | .01 (.86) | .25 (.78)

3. Primary Outcome: Specific Aim 2: Distress Tolerance
Description: Distress Tolerance (DT) assessment includes the Distress Intolerance Index (DII) and the computerized Mirror-Tracing Persistence Task (MTPT-C) which are z-scored and aggregated to form a single DT index.The Distress Tolerance Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched children). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population and with higher scores reflecting worse tolerance.
Time Frame: 1 Week
Population: Statistics are based on all cases with valid data for all variables in the model.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Working Memory Intervention | Control Informational Intervention | Distress Tolerance Intervention
Number analyzed (Participants) | 23 | 27 | 28
z-score | .17 (.80) | .24 (.84) | -.04 (.76)

4. Primary Outcome: Specific Aim 3: Smoking Risk (Standard Smoking Assessment)
Description: The Standard Smoking Assessment is one of 3 assessments of smoking risk along with the B-IAT and the Delay Discounting task. Reported here are the results from the SSA, a 5-item scale asking about attitudes and likelihood of smoking with total scores ranging from 0 (no susceptibility) to 11 (highest susceptibility). The natural log of these scores are reported, with higher scores indicating higher susceptibility.
Time Frame: 1 Week
Population: Statistics are based on all cases with valid data for all variables in the model.
Measure: Mean (Standard Deviation); unit: natural log of units on a scale
Arm/Group | Working Memory Intervention | Control Informational Intervention | Distress Tolerance Intervention
Number analyzed (Participants) | 19 | 22 | 23
natural log of units on a scale | .25 (.50) | .29 (.55) | .31 (.46)

5. Primary Outcome: Specific Aim 3: Smoking Risk (B-IAT)
Description: The brief Implicit Attitudes Test is one of 3 assessments of smoking risk along with the Delay Discounting task and the SSA. Reported here are the d-scores from the B-IAT task. Participants sorted stimuli into "positive" or "negative" categories in 4 blocks--2 of which included "Smoking" and "I feel positive," the other 2 including "Smoking" and "I feel negative." Shorter response times when sorting "Smoking--Positive" versus "Smoking--Negative" blocks indicate implicit tendency to associate "smoking" with "positive." Standardized difference scores (d-scores) were computed using the improved scoring algorithm recommended by prior research (Greenwald, Banaji, & Nosek, 2003). Higher d-scores indicate less positive implicit attitudes towards smoking.
Time Frame: 1 Week
Population: Statistics are based on all cases with valid data for all variables in the model.
Measure: Mean (Standard Deviation); unit: Standardized Difference Scores
Arm/Group | Working Memory Intervention | Control Informational Intervention | Distress Tolerance Intervention
Number analyzed (Participants) | 22 | 26 | 27
Standardized Difference Scores | .19 (.62) | .24 (.32) | .16 (.46)

6. Primary Outcome: Specific Aim 3: Smoking Risk (Delay Discounting Task)
Description: The Delay Discounting task is one of 3 assessments of smoking risk along with the B-IAT and SSA. It includes a series of computerized decisions in which participants select a money award immediately or a larger award in 7, 14, or 30 days time. Participants were notified that they would be paid the amount selected on one randomly selected trial. K-values were submitted for analyses with higher scores representing great discounting of delayed rewards, meaning that higher scores reflect greater tendency to select the immediate award. Natural logs of K-values were used if K-values showed a large amount of skew. Reported here are the natural logs of k-values from the delay discounting task. Natural logs are used to reduce skew of k-values.
Time Frame: 1 Week
Population: Statistics are based on all cases with valid data for all variables in the model.
Measure: Mean (Standard Deviation); unit: natural log of k-values
Arm/Group | Working Memory Intervention | Control Informational Intervention | Distress Tolerance Intervention
Number analyzed (Participants) | 23 | 26 | 28
natural log of k-values | -2.95 (2.78) | -3.69 (2.30) | -3.27 (2.40)

7. Primary Outcome: Specific Aim 4: Actual Smoking Status
Description: The piCO Smokerlyzer is a tool used to assess amount of carbon monoxide exhaled by a participant, with scores ranging from 0 to 150 parts per million (PPM), with scores under 3 indicating non-smoking and scores over 36 indicating very heavy addiction. The Timeline Follow Back is a self-report measure in which participants report the amount of cigarettes smoked each day for the last month. Mean proportions of smokers are reported (0=no smoking, 1=smoking) with smoking behaviors assessed via the piCO Smokerlyzer and the Timeline Follow Back.
Time Frame: 1 Week
Population: Statistics are based on all cases with valid data for all variables in the model.
Measure: Mean (Standard Deviation); unit: Proportion of Smokers
Arm/Group | Working Memory Intervention | Control Informational Intervention | Distress Tolerance Intervention
Number analyzed (Participants) | 20 | 21 | 25
Proportion of Smokers | .10 (.31) | .00 (.00) | .08 (.28)

ADVERSE EVENTS:
Time Frame: 1 Week
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Distress Tolerance Intervention | Working Memory Intervention | Control Informational Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-06-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT03058991/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03058991/SAP_001.pdf